CLINICAL TRIAL: NCT01652209
Title: A Randomized,Open labEled, muLticenter Trial for Safety and Efficacy of Intracoronary Adult Human Mesenchymal stEm Cells Acute Myocardial inFarction
Brief Title: To Evaluate the Efficacy and Safety of Hearticelgram®-AMI in Patients With Acute Myocardial Infarction.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMC-BD-CT-P-003
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): After implementing PCI, contemporary drug treatment is conducted.
  *Contemporary drug treatment is a general drug treatment (Unfractionated heparin, Low Molecular Weight Heparin, Glycoprotein llb/llla inhibitor, Aspirin, clopidogrel or Ticlopidine, Nitrate, ACE inhibitor or ARB, β-blocker, CCB, Diuretics, Statin, etc.)
- Single dose of Hearticellgram-AMI (Experimental): Within 30 days (+ / -7 days) after aspirating bone-marrow, approximately 1×10^6/kg (refer to usage/dosage according to mass) of autologous bone marrow-derived mesenchymal stem cells are adminstered into the infarct coronary artery using balloon tipped catheter. Furthermore, contemporary drug treatment is conducted.
  Interventions: Biological: Hearticellgram-AMI

INTERVENTIONS:
Biological: Hearticellgram-AMI
  Other Names: (Autologous bone marrow derived mesenchymal stem cells)
  Arms: Single dose of Hearticellgram-AMI

SUMMARY:
Through the injection of Hearticellgram-AMI into acute myocardial infarction patients who are the primary targets of the drug, long term efficacy in the improvement of the left ventricle ejection fraction upon the first cell treatment is to be evaluated and compared with the current existing treatments (contemporary drug treatment).

This study will also compare the efficacy and safety of single dose of hearticellgram-AMI.

DETAILED DESCRIPTION:
We are enrolling a patient who had successful conventional percutaneous coronary intervention after acute myocardial infarction. Patients are allocated to one of three groups (group1=comparator, group2= one dose of hearticellgram-AMI).

single dose of hearticellgram-AMI have been attained new drug approval from MFDS (related to NCT01392105).

ELIGIBILITY:
Inclusion Criteria:

1. As of the date of written consent, between 20 and 75 years of age
2. Those with less than 50% of the left ventricular ejection fraction (LVEF) on echocardiography performed after percutaneous coronary intervention (PCI) (evaluated by investigator)
3. Who has been identified as an acute myocardial infarction in any of the following on an electrocardiogram (12-lead electrocardiography, ECG) performed before PCI

   * ST-segment elevation 0.1 mV in two or more limb leads or
   * 0.2 mV elevation in two or more contiguous precordial leads indicative of acute myocardial infarction (AMI)
4. Those identified as anterior wall MI
5. Who meet the above criteria and have successfully reperfused within 72 hours after the onset of chest pain
6. Who can conduct clinical trials according to the clinical trial protocol
7. Who has consented in writing to voluntarily participate in this clinical trial (owner or legal representative)

Exclusion Criteria:

1. Who have not been diagnosed with malignant blood diseases (acute myelogenous leukemia, acute lymphocytic leukemia, non-Hodgkins lymphoma, Hodgkins lymphoma, multiple myelopathy) within 5 years of screening criteria
2. Patients with severe aplastic anemia
3. Patients with solid cancers in their previous medical history (within 5 years)
4. Patients whose blood serum AST/ASL rates are more than three times the normal maximum rate, and whose creatinine rates are more than 1.5 times the normal maximum rate (but AST in myocardial infarction patients can temporarily rise, thus, as decided by the researchers, if there is no damage to the liver function, the rise will not be taken into consideration)
5. Patients who have implemented Coronary Artery Bypass Graft(CABG)
6. Patients with chronic heart failure (patients with medical history of heart failure medical history at least three months before the occurrence of acute myocardial infarction)
7. Patients who cannot proceed with cardiac catheterization
8. Patients who had been continuously taking large doses of steroids (1mg/kg/day) or antibiotics for severe infections from one month prior to registration
9. Patients who had major surgical operations, organ biopsy, or significant external injury as determined by the researcher, within three months before registration
10. Patients who have head injuries or other external injuries after the development of myocardial infarction
11. patients with stroke or transient ischemic attack within six months before registration, patients with history of central nervous system disease (tumor, aneurysm, brain surgery etc.)
12. Patients with low survival ability after cardiopulmonary resuscitation within last 2 weeks.
13. Patients with positive for HIV, HBV, HCV, Syphilis
14. pregnant women or likely to be pregnant or lactating women
15. Patients with drug abuser within last 1 year.
16. Patients with participating other clinical trials with last 1 month.
17. When the possibility of tumor occurrence is seen when the tester judges even one of the tumor marker tests during screening
18. Who are judged to be inappropriate to participate in this test when judged by the examiner

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
LVEF amount of change | 13 months after the cell treatment
  Left ventricle ejection fraction (LVEF) measured 13 months after the cell treatment (MRI measurement)

SECONDARY OUTCOMES:
LVEF amount of change | 6 months after the cell treatment
  Left ventricle ejection fraction (LVEF) measured 6 months after the cell treatment (MRI measurement)
Infarct size amount of change | 6, 13 months after the cell treatment
  Change in infarct size evaluated by MRI at 6 and 13 months compared to before administration
Left ventricle end systolic size change | 6, 13 months after the cell treatment
  Change in left ventricular end systolic size evaluated by MRI at 6 months and 13 months compared to before administration
Left ventricular end-diastolic size change | 6, 13 months after the cell treatment
  Change in left ventricular end diastolic size evaluated by MRI at 6 months and 13 months compared to before administration
Incidence of critical heart events | Within 24 months after the cell treatment
  The incidence of major cardiac events (death, hospitalization for cardiac shock or heart failure, recurrence of myocardial infarction, occurrence of severe arrhythmias) within 24 months after administration
Heart rate variability change amount | 13 months after the cell treatment
  Heart rate variability change at 13 months compared to before administration (24 hours Holter measurement)
Left ventricular local wall movement disorder index change | 6, 13 months after the cell treatment
  The amount of change in the left ventricular local wall movement impairment index evaluated by echocardiography at 6 and 13 months compared to before administration
N-terminal pro-brain natriuretic peptide (NT-proBNP) change | 6, 13 months after the cell treatment
  Changes in N-terminal pro-brain natriuretic peptide (NT-proBNP) at 6 and 13 months compared to before administration

CONTACTS AND LOCATIONS:
Overall Officials: Jeonghan Yoon, Ph.D. M.D., Principal Investigator — Wonju Severance Christian Hospital
Locations (10):
- South Korea (10):
  - Kangwon National University Hospital, Chuncheon
  - Chonnam National University Hospital, Gwangju
  - Yongin Severance Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Chungnam National University Hospital, Jungnam
  - Catholic University of Korea, Seoul ST. Mary's Hospital., Seoul
  - Korea University Medicine, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Seoul
  - Wonju Severance Christian Hospital, Wŏnju